CLINICAL TRIAL: NCT04842825
Title: A Randomized Controlled Study on Sequential Therapy of Kidney Tonifying and Blood Regulating Herbs to Improve the Success Rate of IVF-ET in Patients With Ovarian Reserve Dysfunction
Brief Title: Sequential Therapy of TCM Herbs to Improve the Success Rate of IVF-ET in Diminished Ovarian Reserve Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00006761-M2020368
Record Dates: First submitted 2021-03-17; First posted 2021-04-13 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Infertility, Female
Keywords: infertility; traditional chinese medicine; ovarian reserve; Fertilization in Vitro; Embryo Transfer
MeSH Terms: conditions — Infertility, Female; Infertility | interventions — si-wu-tang; Injections

STUDY DESIGN:
Intervention Model Description: To further investigate its role in improving pregnancy outcomes of IVF-ET in diminished ovarian reserve (DOR) infertility, in this randomized, controlled clinical trial, 200 patients with DOR infertility who intended to undergo IVF-ET will be randomly divided into two groups: a treatment group (Western conventional treatment + kidney-tonifying and blood-regulating herbs) and a control group (Western treatment only). The intervention will be started from the 5th day of menstruation for two menstrual cycles before undergoing IVF-ET until 14 days after transfer.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kidney-tonifying and blood-regulating herbs treatment group (Experimental): the treatment group will receive sequential treatment with the Chinese herbal formula for tonifying the kidney, nourishing the blood, and activating the blood 2 months before the proposed ET to regulate menstruation and improve ovarian reserve function. Treatment with the Chinese herbal formula will continue on the 5th day of menstruation after entering the super-ovulation cycle.
  Interventions: Drug: Er Zhi Wan combined with Si Wu Tang
- Western medicine group (Active Comparator): The control group will be treated with conventional Western medicine
  Interventions: Drug: Recombinant Human Follitropin Alfa 、Fructose 、Tetyacycline Hydrochloride Capsules、Cetrorelix Acetate Powder

INTERVENTIONS:
Drug: Er Zhi Wan combined with Si Wu Tang — The TCM medicines used will be Radix et Rhizoma Ligustrum 15 g, Radix Morindae Sinensis 12 g, Fructus Lycii 15 g, Semen Cuscutae 20 g, Radix Rehmanniae 20 g, Radix Angelicae Sinensis 10 g, Radix Paeoniae Alba 12 g, Radix Yam 20 g. The hospital will be responsible for the decoction of 200 mL per dose, 1 dose per day, divided into 2 doses in the morning and in the evening, for 10-15 days. According to follicular development and endometrial growth monitored by ultrasound, the herbs will be changed to Curculus 10 g, Xianling spleen 15 g, Morinda officinalis 15 g, Cuscutae 20 g, Amethyst 15 g, Rehmannia 20 g, Angelica 15 g, Chuanxiong 10 g，which will be taken for 10-15days.
  After ET, the treatment group will continue to take Chinese herbal medicine, changing to Cuscuta 15 g, Sambucus 15 g, Chuan Guan Gong 10 g, Agaricus 9 g, Shu Di 15 g, Angelica 10 g, Bai Shao 12 g for 14 days
  Other Names: conventional western medicine(Recombinant Human Follitropin Alfa for Injection、Fructose Injection、Tetyacycline Hydrochloride Capsules、Cetrorelix Acetate Powder for Injection )
  Arms: kidney-tonifying and blood-regulating herbs treatment group
Drug: Recombinant Human Follitropin Alfa 、Fructose 、Tetyacycline Hydrochloride Capsules、Cetrorelix Acetate Powder — The control group will be treated with conventional Western medicine（The specific drug dose is determined according to the individual level of patients）
  Other Names: (Recombinant Human Follitropin Alfa for Injection、Fructose Injection、Tetyacycline Hydrochloride Capsules、Cetrorelix Acetate Powder for Injection )
  Arms: Western medicine group

SUMMARY:
In the early stage, our team found that traditional Chinese medicine (TCM) intervention aimed at Nourishing kidney and regulating blood circulation in vitro fertilization and embryo transfer(IVF-ET) can improve the clinical pregnancy rate. In order to further study the role of TCM in improving the pregnancy outcome of IVF-ET in infertility due to decreased ovarian reserve (DOR). A randomized controlled clinical trial was used in this study. 200 infertile patients with DOR were randomly divided into two groups. The control group was treated with conventional modern medicine, and the treatment group was treated with traditional Chinese herbs on the basis of conventional modern medicine.

The intervention started from the 5th day of the first menstrual cycles after enrollment and lasted for three months before IVF-ET. After the transplantation, the TCM treatment continues for 14 days. The number of oocytes, antral follicles, anti-Mullerian hormone(AMH), serum follicle-stimulating hormone(FSH), and clinical pregnancy rate will be observed to evaluate the effect of traditional Chinese medicine on the improvement of ovarian function, pregnancy outcome, and fertility of DOR patients.

DETAILED DESCRIPTION:
The study will be conducted on patients with DOR attending our reproductive medicine centre for proposed IVF-ET between January 2021and December 2022.

The trial is designed as a randomised, controlled clinical trial with two groups established by 1:1 equal allocation, a treatment group with interventions using herbs to tonify the kidneys and regulate blood and a control group treated using conventional Western medicine.

Random numbers will be prepared by an independent third-party statistician who prepared a list of random group codes for this study. Enrolled subjects will be given a subject number during the screening process and, upon formal enrolment, will be randomly assigned to either the test or control group with a corresponding random number.

Treatment method Phase I: The control group will be treated with conventional Western medicine, whereas the treatment group will receive sequential treatment with the Chinese herbal formula 2 months before the proposed embryo transfer(ET) to regulate menstruation and improve ovarian reserve function. Treatment with the Chinese herbal formula will start on the 5th day of menstruation after entering the super-ovulation cycle. The medicines used will be Er Zhi Wan combined with Si Wu Tang (Radix et Rhizoma Ligustrum 15 g, Radix Morindae Sinensis 12 g, Fructus Lycii 15 g, Semen Cuscutae 20 g, Radix Rehmanniae 20 g, Radix Angelicae Sinensis 10 g, Radix Paeoniae Alba 12 g, Radix Yam 20 g); which will be taken for 10-15days. After ovulation, the herbs used to warm the kidney and regulate the blood will be changed to Er Xian Promoting Pregnancy Decoction with Si Wu Decoction (Curculus 10 g, Xianling spleen 15 g, Morinda officinalis 15 g, Cuscutae 20 g, Amethyst 15 g, Rehmannia 20 g, Angelica 15 g, Chuanxiong 10 g); which will be taken for 10-15days. The hospital will be responsible for the decoction of 200 mL per dose, 1 dose per day, divided into 2 doses in the morning and in the evening.

Phase 2: After ET, the control group will be treated conventionally with no TCM intervention, and the treatment group will continue to take Chinese herbal medicine, changing to tonifying the kidney, regulating blood, and calming the foetus, using Shou Foetus pill combined with Si WuTang with addition and subtraction (Cuscuta 15 g, Sambucus 15 g, Chuan Guan Gong 10 g, Agaricus 9 g, Shu Di 15 g, Angelica 10 g, Bai Shao 12 g), which will be taken until the 14th day of transplantation.

Medication Patients that meet the inclusion criteria will be assigned to one of two groups according to a randomisation table after completing the relevant tests and signing the informed consent form. The control group will be treated routinely, and the treatment group will begin taking the assigned drugs on the 5th day (with no intervention drugs taken on days 1-4) of menstruation for two menstrual cycles before IVF until the day of ET and then continue the intervention for 14 days after ET.

Follow-up plan Blood tests to measure progesterone and human chorionic gonadotropin(hCG) will be performed 14 days after fresh or frozen ET. If the blood results confirm pregnancy, a clinical pregnancy will be confirmed after 2 weeks by vaginal ultrasound. When a gestational sac is seen in the uterus, the presence or absence of ectopic pregnancy and the number of implanted foetuses will be determined. Those with clinical pregnancy will be followed for final pregnancy outcome (miscarriage/live birth, week of delivery, and a number of new-borns), delivery (mode of delivery and pregnancy complications), and offspring (sex, weight, length, presence of birth defects, and stillbirth). Follow-up will be limited to subjects with transferred embryos obtained from egg retrieval in this study. In the case of subject withdrawal or dropout from the study, detailed reasons will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Consent to participate in this clinical trial and sign an informed consent form.
2. Age ≤40 years, regular menstrual cycle between 21and 35 days in length.
3. Meet the Western diagnostic criteria for DOR.
4. Meet the criteria for identifying kidney deficiency in Chinese medicine.
5. Planning to undergo IVF-ET for pregnancy.

Exclusion Criteria:

1. History of two or more previous spontaneous abortions (excluding biochemical pregnancy abortions) or three or more previous ETs without obtaining a clinical pregnancy.
2. Premature ovarian failure or ovarian gonadotropin resistance syndrome.
3. Untreated uterine anomalies or abnormalities, including double uterus or longitudinal uterus (complete or incomplete).
4. Untreated hydrocele on one or both fallopian tubes (confirmed by hysterosalpingography).
5. Uterine adhesions, endometriosis, adenomyosis, endometrial lesions (submucosal fibroids, endometrial polyps, etc.), or uterine fibroids >4 cm.
6. Endocrine disorder affecting ovulation, such as polycystic ovary syndrome, hyperprolactinaemia, hyperandrogenaemia, hypothyroidism, or adrenal abnormalities.
7. Infertility with abnormal ovarian function due to immune factors, genetic factors, or congenital physical defects.
8. Previous pelvic radiotherapy.
9. Known or suspected sex hormone-related malignancy.
10. Allergy to or intolerance of the drugs used in the study.
11. Combined contraindications to assisted reproductive technology or pregnancy, such as uncontrolled abnormalities of liver and kidney function, diabetes mellitus (glycosylated haemoglobin ≤7%, fasting blood glucose <10 mmol/L ), hypertension, thyroid disease, symptomatic heart disease, moderate to severe anaemia, history of malignancy or thromboembolism or propensity to thrombosis, severe psychiatric disorder, acute infections of the genitourinary system, sexually transmitted diseases, serious adverse habits such as drug abuse, exposure to teratogenic amounts of radiation, toxins, or drugs (such as prednisone or other hormones, adrenaline, antibiotics, or hypertension, cardiovascular, or antiviral medications) during the active procedure period , and uterine factor infertility or physical illness which prevents the ability to bear a pregnancy.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of eggs obtained | up to 15 weeks from enrollment
  Obtained by blood sampling before the proposed IVF-ET
Change from Baseline concentration of Serum anti-Mullerian hormone(AMH) before the proposed IVF-ET | The 5th day of menstruation in the month of enrollment and Before the proposed IVF-ET（up to 15 weeks from the enrollment）
  Obtained by blood sampling before taking TCM herbs and before the proposed IVF-ET
Change from Baseline concentration of Serum follicle-stimulating hormone (FSH) before the proposed IVF-ET | The 5th day of menstruation in the month of enrollment and Before the proposed IVF-ET（up to 15 weeks from the enrollment）
  Obtained by blood sampling before taking TCM herbs and before the proposed IVF-ET
Clinical pregnancy rate (%): number of clinical pregnancies/total number of ET cycles | up to 19 weeks from the enrollment
  Follow up by telephone calls 30days after the IVF-ET

SECONDARY OUTCOMES:
Change from Baseline concentration of antral follicle count(AFC) before the proposed IVF-ET | The 5th day of menstruation in the month of enrollment and Before the proposed IVF-ET（up to 15 weeks from the enrollment）
  Obtained by blood sampling before taking TCM herbs and before the proposed IVF-ET
Concentration of follicular E2 level on the day of human chorionic gonadotropin(hCG) injection | up to 15 weeks from enrollment
  Obtained by blood sampling before the proposed IVF-ET
Change from Baseline concentration of Serum luteinising hormone(LH) before the proposed IVF-ET | The 5th day of menstruation in the month of enrollment and Before the proposed IVF-ET（up to 15 weeks from the enrollment）
  Obtained by blood sampling before taking TCM herbs and before the proposed IVF-ET
Quality egg rate (%) | up to 15 weeks from enrollment
  Before the proposed IVF-ET
Total amount of ovulation-promoting drugs | up to 15 weeks from enrollment
  Before the proposed IVF-ET
Fertilisation rate (%) | up to 15 weeks from enrollment
  Before the proposed IVF-ET
Implantation rate (%): number of gestational sacs/number of embryos transferred | up to 19 weeks from the enrollment
  30days after the IVF-ET
Concentration of human chorionic gonadotropin(hCG) | up to 17 weeks from the enrollment
  14days after the IVF-ET
Concentration of progesterone | up to 17 weeks from the enrollment
  14days after the IVF-ET

CONTACTS AND LOCATIONS:
Overall Officials: Dong Li, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China, China

IPD SHARING:
Plan to Share IPD: No